CLINICAL TRIAL: NCT00482586
Title: Outcomes Following Image-Guided Therapy for Hepatic Malignancies
Brief Title: Quality of Life in Patients With Liver Cancer Treated With Image-Guided Therapy
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Meranze, Professor of Radiology, Vanderbilt University
Other Study IDs: CDR0000546520; P30CA068485 (NIH); VU-VICC-GI-0372 (Other: Vanderbilt University); VU-VICC-IRB-020874 (Other: Vanderbilt University)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: adult primary liver cancer; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Embolization, Therapeutic; Chemoembolization, Therapeutic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Image-guided Therapy: Patients undergoing Image-guided Therapy of Hepatic Neoplasms.
  Interventions: Other: medical chart review; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: medical chart review — Review the medical charts of patients with hepatic neoplasms who undergo Image-guided Therapy.
  Other Names: Ablation; Embolization
Other: questionnaire administration — Patients with hepatic neoplasms who undergo Image-guided Therapy
  Other Names: Ablation; Embolization; Chemo-embolization
Procedure: quality-of-life assessment — Patients with hepatic neoplasms who undergo Image-guided Therapy
  Other Names: Ablation; Embolization; Chemoembolization

SUMMARY:
RATIONALE: Gathering information about quality of life over time from patients with liver cancer treated with image-guided therapy may help the study of cancer in the future.

PURPOSE: This clinical trial is gathering information about quality of life over time from patients with liver cancer treated with image-guided therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop a data repository for clinical and health-related quality of life outcome measures in patients with hepatic malignancies treated with image-guided therapies.

OUTLINE: This is a pilot, prospective, longitudinal study.

Patients complete a standard questionnaire assessing health-related quality of life at baseline, during routine follow-up care after image-guided therapy, and then annually thereafter. Health and disease status and the development of other illnesses are assessed by medical record review.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing concurrent image-guided therapy for hepatic malignancies using any of the following imaging techniques:

  * X-ray
  * Ultrasound
  * MRI
  * CT scan
  * Nuclear medicine imaging

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic neoplasms who undergo Image-guided Therapy
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2003-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Development of a data repository for clinical outcome measures by conducting a medical record review at baseline, during routine follow-up after image-guided therapy, and then annually thereafter | one year
Development of a data repository for health-related quality of life outcome measures by administering the Medical Outcomes Study Short Form questionnaire at baseline, during routine follow-up after image-guided therapy, and then annually thereafter | one year

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Meranze, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee